CLINICAL TRIAL: NCT06127667
Title: Brain Vascular and Neural Function Linked to Balance Across the Adult Lifespan
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PT-2023-32375
Record Dates: First submitted 2023-10-29; First posted 2023-11-13 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Neurotypical; Cognitively Normal
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Healthy participants in 3 age groups
  Interventions: Behavioral: aerobic exercise

INTERVENTIONS:
Behavioral: aerobic exercise — use of single bout of aerobic exercise

SUMMARY:
This is a single-arm, two-visit, non-randomized, cross sectional study identified as an intervention due to the use of a single bout of aerobic exercise to assess cerebrovascular function under the NIH rules. This study is not masked and its primary purpose is to develop a basic science understanding of the relationship between cerebrovascular health and balance control with aging. This study will involve 102 individuals classified as younger adults, middle-aged adults, and older adults who are neurotypical and cognitively normal. The primary outcome from a clinical trials perspective will be cerebrovascular response to a bout of aerobic exercise (i.e. change in cerebral blood flow with the performance of aerobic exercise on a recumbent stepper exercise machine). Non-interventional outcomes will be EEG measures of cortical activity and biomechanical kinetic and kinematic data recorded during standing balance reactions, as well as biological blood samples for genomic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age within the following 3 group age ranges, 21-30yo; middle-aged: 40-55yo; older: 65-95yo adults
* the absence of major orthopedic disability
* cognitively normal (MoCA score ≥ 26/30 in older adult group)
* vision that is 20/40 or better with or without corrective lenses, (5) the ability to consent and communicate with researchers
* English speaking
* ability to stand for 3 minutes and walk 10 meters with or without an assistive device and without the assistance of another person.

Exclusion Criteria:

* insulin-dependent diabetes
* peripheral neuropathy
* myocardial infarction or symptoms of coronary artery disease within 2 years
* congestive heart failure or class IV heart failure
* any significant sensory impairment affecting balance or cognition; visual, vestibular, or auditory impairments.

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
cerebral blood flow velocity assessed using transcranial Doppler ultrasound | 1 week
  Includes recordings from transcranial Doppler ultrasound of cerebral blood flow (CBF) velocity performed at the first session during rest, sit-to-stand, transfer, and single bout of aerobic exercise.
Kinetic center of pressure rate of rise post-balance perturbation, assessed biomechanically. | 1 week
  Recordings from 64-channels of EEG electrodes, kinetic, and kinematic biomechanical data during standing balance reactions will be collected.
Prefrontal-M1 coherence an S1-M1 coherence post-balance perturbation, assessed using EEG | 1 week
  Recordings from 64-channels of EEG electrodes, kinetic, and kinematic biomechanical data during standing balance reactions will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Palmer, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States